CLINICAL TRIAL: NCT04965064
Title: An Open-Label Phase II Trial of Neratinib Plus Capecitabine in Subjects With HER2-Negative Metastatic Breast Cancer With Brain Metastases and Abnormally Active HER2 Signaling
Brief Title: Trial of Neratinib Plus Capecitabine in Subjects With HER2-Negative Metastatic Breast Cancer With Brain Metastases and Abnormally Active HER2 Signaling
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Ajay Dhakal, Assistant Professor - Department of Medicine , Hematology/Oncology (SMD), University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UBRS20139
Record Dates: First submitted 2021-07-02; First posted 2021-07-16 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer
Keywords: HER2-negative metastatic breast cancer; Brain metastases
MeSH Terms: conditions — Breast Neoplasms; Brain Neoplasms | interventions — Capecitabine; neratinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Experimental: Capecitabine and Neratinib. (Experimental): Neratinib 240 mg PO QD Daily On-going
  Capecitabine 750 mg/m2 PO bid Days 1-14, 7 days off On-going
  Interventions: Drug: Capecitabine and Neratinib.

INTERVENTIONS:
Drug: Capecitabine and Neratinib. — Neratinib 240 mg PO QD Daily On-going Capecitabine 750 mg/m2 PO bid Days 1-14, 7 days off On-going

SUMMARY:
The purpose of this research is to look at the safety and effectiveness of a HER2-targeted therapy neratinib when given with capecitabine, a chemotherapy, for breast cancer patients with brain metastases whose tumors were HER2-negative by standard tests but showed abnormal HER2 activity based on the CELsignia results.

DETAILED DESCRIPTION:
The purpose of this research is to look at the safety and effectiveness of a HER2-targeted therapy neratinib when given with capecitabine, a chemotherapy, for breast cancer patients with brain metastases whose tumors were HER2-negative by standard tests but showed abnormal HER2 activity based on the CELsignia results. The CELsignia test results might predict whether this breast cancer type will respond to treatment with neratinib and capecitabine.

Neratinib is called a HER2-targeted therapy because it stops cancer cells from growing by targeting and blocking the HER2 proteins that help cancer cells grow. Neratinib is an oral drug approved by the U.S. Food and Drug Administration (FDA) to treat HER2-positive breast cancer. It is considered investigational in this study because your breast cancer was determined to be HER2-negative by the standard method of testing. However, the CELsignia test showed that your breast cancer cells have HER2 pathway activity that might respond to HER2-targeted treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet all of the following criteria to be enrolled:

  * Male/Female
  * At least 18 years of age
  * Histologically confirmed HER2 negative breast cancer determined from the most recent tumor sample (primary or metastatic), as per the current American Society of Clinical Oncology and College of American Pathologists HER2 testing guidelines.
  * For ER positive breast cancer patients: prior treatment with a CDK4/6 inhibitor and endocrine therapy in required in the metastatic settings. If a patient has received a CDK4/6 inhibitor plus endocrine therapy in the adjuvant settings and the cancer recurred while on the CDK4/6 inhibitor or within 12 months of the end of CDK4/6 inhibitor treatment, then the patient will eligible without getting a CDK4/6 inhibitor and endocrine therapy in the metastatic setting.
  * For triple negative breast cancer patients: no specific prior anti-cancer treatment is required.
  * Have radiological evidence of one or more brain metastases.
  * Ability to obtain an MRI.
  * Has a radiological evidence of a measurable disease (per RECIST 1.1) outside of the brain which is accessible to a biopsy
  * Willing to undergo a research core biopsy of the tumor tissue
  * Considered to be medically fit for undergoing a biopsy
  * Subjects anticipated by the investigator to be a candidate for systemic therapy immediately or in the future.
  * Ability to understand the investigational nature of the study and sign the informed consent
* Key Criteria for Step 1 Registration:

  * Abnormally active HER2 signaling as determined by the CELsignia test on the tumor tissue.
  * New or progressive brain metastases defined as any one of the following:
  * Untreated measurable lesions in patients who have received surgery and/or stereotactic radiosurgery (SRS) to one or more other lesions.
  * Residual or progressive lesions after surgery if asymptomatic.
  * Patients who have had prior whole-brain radiotherapy (WBRT) and/or SRS and then whose lesions have progressed by RANO-BM criteria or there are new lesions are eligible. Lesions treated with SRS may be eligible if there is unequivocal evidence of progression.
  * Patients who have not previously been treated with cranial radiation (e.g., WBRT or SRS) are eligible, but such patients must be asymptomatic and neurologically stable from their CNS metastases.
  * Measurable brain metastases with at least one lesion > 5 mm in longest diameter AND is/are new or progressive lesion/s as defined by criterion B.
  * Ability to obtain MRI
  * No major surgery within 10 days prior to registration. Surgeries should be avoided any time after registration during the study treatment, but minor procedures like dental extractions and surgeries deemed important to maintain or improve patients' quality of life and are allowed.
  * A minimum of 14 days since the last dose of chemotherapy except for the optional pre-Step 1 capecitabine. If pre-step 1 optional capecitabine was administered, then a minimum of 7 days from the last dose of Capecitabine is required before registration. There is no limit on the number of previous chemotherapy regimens for eligibility.
  * A minimum of 7 days since the last dose of any hormonal therapy (no limit on the number of previous hormonal regimens for eligibility) except fulvestrant. A minimum of 28 days since the last dose of fulvestrant before registration.
  * A minimum of 21 days since the last dose of targeted therapy (e.g., a CDK4/6 inhibitor, PI3kinase inhibitors, etc.)
  * A minimum of 7 days since the last fraction of extracranial radiation and has recovered from any acute toxic effects of radiation therapy
  * A minimum of 30 days since the last dose of any investigational cancer treatment or any immunotherapy
  * ECOG performance status of 0 -2
  * Left ventricular ejection fraction ≥ 50% at baseline
  * Prior treatment-related major organ toxicities recovered to ≤grade 1
  * Adequate bone marrow, hepatic, renal, and coagulation function
  * Post-menopausal, surgically sterile, or willing to use a reliable form of contraception while on the study and for 180 days after discontinuing either study treatment. The patients that can father children are willing to use highly effective contraception for at least 90 days following last dose of either study treatment.
  * Ability to understand the investigational nature of the study and sign the informed consent

Exclusion Criteria:

* Subjects must NOT meet any of the following criteria to be enrolled:

  * Patients who have received capecitabine for the treatment of the current breast cancer in the metastatic setting
  * Patients who have received capecitabine only in the perioperative setting for the primary early-stage breast cancer AND the breast cancer recurred while taking capecitabine or within 180 days of the last dose of capecitabine therapy.
  * History of other malignancies other than the following: 1. adequately treated non-melanoma skin cancer, 2. curatively treated in-situ cancer of the cervix 3. other solid tumors which have been curatively treated AND no evidence of recurrence in the last 2 years.
  * Gastrointestinal tract disease resulting in an inability to absorb oral medication
  * Known hypersensitivity to the study drugs or their components
  * Pregnant or breast-feeding
  * Known or suspected leptomeningeal disease
  * Known bleeding or coagulation issues, subject taking anticoagulants or having bleeding diathesis that may significantly increase the risk of bleeding during the biopsy. If the subject is on anticoagulation, perioperative management of anticoagulation should be done per institutional practice.
  * Chronic and concomitant use of strong or moderate CYP3A4 inhibitors and strong or moderate CYP3A4 inducers. These drugs should be stopped at least 14 days prior to registration to Step 0.
  * Current uncontrolled medical conditions that could limit a subject's ability to undertake study therapy
  * Inflammatory bowel disease with diarrhea as a major component
* Key Criteria for Step 1:

Subjects must NOT meet any of the following criteria to be enrolled:

* Normally active HER2 signaling as determined by the CELsignia test on the tumor tissue
* Inconclusive HER2 signaling testing by the CELsignia test on the tumor tissue
* Whole-brain radiotherapy in the prior three months
* Resting blood pressure higher than systolic of 160 and/or diastolic of 110 mmHg or poorly controlled hypertension, history of labile hypertension, or poor compliance with anti-hypertensive medication
* Serious cardiac illness or condition including, but not limited to, clinically significant congestive heart failure, high-risk uncontrolled arrhythmias, unstable angina pectoris requiring medication, or clinically significant valvular heart disease
* History of pulmonary embolus or deep vein thrombosis diagnosed within the previous three months
* Current uncontrolled medical conditions that could limit a subject's ability to undertake study therapy
* Known or suspected leptomeningeal disease
* Inflammatory bowel disease with diarrhea as a major component
* Chronic and concomitant use of strong or moderate CYP3A4 inhibitors and strong or moderate CYP3A4 inducers. These drugs should be stopped at least 14 days prior to registration to Step 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2022-09-23 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
overall survival | 24 months
  The study will assess how long participants with HER2 negative metastatic breast cancer with brain metastasis and abnormal HER2 signalling will survive if treated with capecitabine and neratinib
CNS progression free survival | 24 months
  The study will assess how long participants with HER2 negative metastatic breast cancer with brain metastasis and abnormal HER2 signalling will survive and also not have the cancer get worse in the brain while treated with capecitabine and neratinib

CONTACTS AND LOCATIONS:
Overall Officials: Ajay Dhakal, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided